CLINICAL TRIAL: NCT07219277
Title: Clinical Validation of Early Detection Blood Test for Universal Large-scale Breast Cancer Screening to Improve Early Diagnosis for Women of All Social and Ethnic Backgrounds
Brief Title: Clinical Validation of Early Detection Blood Test for Universal Large-scale Breast Cancer Screening
Status: Not yet recruiting | Type: Observational
Sponsor: Syantra Inc. (Industry)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: SY-2024-01; HT94252410228 (Other Grant/Funding Number: The Assistant Secretary of Defense for Health Affairs)
Record Dates: First submitted 2025-10-15; First posted 2025-10-21 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer, Liquid Biopsy, Early Detection
Keywords: Breast cancer detection; Breast Cancer Screening; Blood Test; Early Detection
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood collection into PAXGene blood RNA tubes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Elevated risk population - Asymptomatic: Women at elevated risk undergoing screening for breast cancer who are currently undergoing asymptomatic screening. Presentation of factor(s) indicating elevated risk for breast cancer development including: germline genetic mutations known to increase risk of breast cancer, very dense (D) breast tissue, family history, and/or clinical risk assessment and scoring at elevated risk (20% or greater lifetime risk, or 3% or greater 10-year risk assessed at age 40, using the Tyrer-Cuzick model (v.7 or v.8) or 1.67% or greater 5-year breast cancer risk using the BCSC model
- Elevated risk population -Recall: Women at elevated risk undergoing screening for breast cancer who are currently undergoing recall screening. Women who have undergone previous MRI and/or screening mammogram or ultrasound indicating follow-up imaging or biopsy recommended and who may have presentation of factor(s) indicating elevated risk for breast cancer development. Factors may include germline genetic mutations known to increase risk of breast cancer, very dense (D) breast tissue, family history, and/or clinical risk assessment and scoring at elevated risk (20% or greater lifetime risk, or 3% or greater 10-year risk assessed at age 40, using the Tyrer-Cuzick model (v.7 or v.8) or BOADICEA v6.0 or 1.67% or greater 5-year breast cancer risk using the BCSC model.
- Recall (Secondary care) Symptomatic population: Women recommended for follow-up due to physical symptoms. This includes recommendation for diagnostic imaging and/or biopsy due to physical symptoms.
- Asymptomatic average, low or unknown risk population: Women undergoing routine screening for breast cancer. Women in the Screening population would have no physical symptoms and be consented near the time of a screening imaging session (within 3 months). Recruitment may also occur after a screening imaging session with a recommendation for follow-up imaging, or after diagnostic imaging with a recommendation for a biopsy as part of the recall population.

SUMMARY:
Breast cancer is the most common cancer that spreads beyond the initial layer of tissue it developed in, and grows into surrounding healthy tissue in women worldwide. It is associated with significant illness and death. Identifying the disease in the early stage is important to achieving positive outcomes in response to diagnosis and treatment.

The Syantra blood test has been developed over the past 10 years. This test involves examining blood samples to identify and analyze specific information. This information is run through a software program that then potentially identifies the presence of breast cancer in the blood sample. This test has the potential to increase early stage detection of breast cancer.

The main goal of this study is to figure out how well the Syantra blood test identifies the presence of breast cancer in women 30-75 years of age. The study will also look at whether things like ethnicity, geography and certain individual characteristics (including breast density and elevated risk of breast cancer development) have an effect on how well the test works.

This study will recruit women who are attending a visit at the site who are aged 30-75 who are undergoing testing for the presence of breast cancer as part of their regular screening or planned follow up imaging and/or biopsy.

Participants who provide consent and meet eligibility criteria will complete a baseline questionnaire and have their blood drawn before any scheduled procedures. Relevant information will be collected from their medical record at the time of joining the study and will be reviewed and updated within 60 days and then again at 12 months following the baseline blood draw. Participants will not have to do anything after the initial visit where they may sign consent, complete the intake questionnaire and have their blood drawn.

DETAILED DESCRIPTION:
Primary Objective: Determine clinical performance metrics of the Syantra blood test in a population of women 30-75 years of age.

Secondary Objectives: Investigate the role of ethnicity, geography, and participant characteristics (including breast density and elevated risk of breast cancer development) on test performance.

Investigate tumor characteristics and test development. Study Design: Non-randomized, blinded, non-interventional, longitudinal, multi-center Investigational Device: Syantra blood test Population: Women age 30-75 years testing for the presence of breast cancer as part of regular breast screening or planned follow-up diagnostic imaging and/or biopsy Accrual Goal: 2,000 women Primary Endpoint: Clinical performance of the Syantra blood test in the primary population Procedure: Participants providing consent and meeting eligibility criteria will complete a baseline questionnaire (demographics and medical history) and have their blood drawn prior to surgical procedure or biopsy (if applicable). Participant medical records will be reviewed to collect relevant history, including imaging studies, surgery, and pathology results, along with medical treatments and patient status.

Follow-up: Medical records for participants will be reviewed and updated after completion of diagnostic procedures (within 60 days) and at 12 months post baseline blood draw to complete recording of procedures and status, including interval cancers or other newly diagnosed diseases. Participants with incomplete records or follow-up will be reviewed annually for imaging, pertinent medical issues, and/or outcomes for up to 5 years.

Biospecimen Retention: De-identified blood samples stored for up to 20 years.

ELIGIBILITY:
1. Elevated risk population sub-group: Women at elevated risk undergoing routine screening for breast cancer.

   A. Asymptomatic Screening Inclusion Criteria
   * Age ≥ 30 and ≤ 75
   * Planned MRI (for women who qualify) and/or planned screening mammogram (and/or breast ultrasound)
   * Presentation of factor(s) indicating elevated risk for breast cancer development

     o Factors may include germline genetic mutations known to increase risk of breast cancer, very dense (D) breast tissue, family history, and/or clinical risk assessment and scoring at elevated risk (20% or greater lifetime risk, or 3% or greater 10-year risk assessed at age 40, using the Tyrer-Cuzick model (v.7 or v.8) or 1.67% or greater 5-year breast cancer risk using the BCSC model
   * Willing and able to give Written Informed Consent and provide a whole blood sample

   Exclusion Criteria
   * Physical breast symptoms or concerns
   * Current or suspected cancer diagnosis
   * Prior BI-RADS 3 or higher imaging results in last 12 months
   * Breast surgery within the previous 12 months (for any reason) or recent breast biopsy (including needle core biopsy) within the last 12 months
   * Previous history of any cancer, except for non-melanoma skin cancer (basal cell carcinoma and squamous cell carcinoma)
   * Previous history of invasive or non-invasive breast cancer
   * Concomitant or other concurrent anti-cancer therapy
   * Blood transfusions within the past 3 months
   * Born biologically male

   B. Recall Inclusion Criteria
   * Age ≥ 30 and ≤ 75
   * Previous MRI (for women who qualify) and/or screening mammogram (and/or breast ultrasound) indicating follow-up imaging or biopsy recommended
   * Presentation of factor(s) indicating elevated risk for breast cancer development

     o Factors may include germline genetic mutations known to increase risk of breast cancer, very dense (D) breast tissue, family history, and/or clinical risk assessment and scoring at elevated risk (20% or greater lifetime risk, or 3% or greater 10-year risk assessed at age 40, using the Tyrer-Cuzick model (v.7 or v.8) or BOADICEA v6.0 or 1.67% or greater 5-year breast cancer risk using the BCSC model.
   * Willing and able to give Written Informed Consent and provide a whole blood sample

   Exclusion Criteria
   * Physical breast symptoms or concerns
   * Breast surgery within the previous 12 months (for any reason) or recent breast biopsy (including needle core biopsy) within the last 12 months
   * Current diagnosis or history of any cancer, including DCIS, with the exception of non-melanoma skin cancer (basal cell carcinoma and squamous cell carcinoma)
   * Blood transfusions within the past 3 months
   * Born biologically male
2. Recall (Secondary care) Symptomatic population: Women recommended for follow-up due to physical symptoms. This includes recommendation for diagnostic imaging and/or biopsy due to physical symptoms.

   Inclusion Criteria
   * Age ≥ 30 and ≤ 75
   * Planned diagnostic breast imaging (mammogram, breast MRI and/or breast ultrasound) and/or breast biopsy, as recall or follow-up from prior examination or to evaluate breast symptom.
   * Willing and able to give Written Informed Consent and provide a whole blood sample.

   Exclusion Criteria
   * Current known cancer diagnosis
   * Breast surgery within the previous 12 months (for any reason) or recent breast biopsy (including needle core biopsy) within the last 12 months
   * History of any cancer, with the exception of non-melanoma skin cancer (basal cell carcinoma and squamous cell carcinoma)
   * Blood transfusions within the past 3 months
   * Born biologically male
3. Asymptomatic average, low or unknown risk population: Women undergoing routine screening for breast cancer. Women in the Screening population would have no physical symptoms and be consented near the time of a screening imaging session (within 3 months). Recruitment may also occur after a screening imaging session with a recommendation for follow-up imaging, or after diagnostic imaging with a recommendation for a biopsy as part of the recall population.

Inclusion Criteria

* Age ≥ 30 and ≤ 75
* Screening mammogram and/or breast ultrasound, breast MRI within 3 months
* Willing and able to give Written Informed Consent and provide a whole blood sample

Exclusion Criteria

* Physical breast symptoms or concerns
* Breast surgery within the previous 12 months (for any reason) or breast biopsy (including needle core biopsy) within the last 12 months
* History of any cancer, including DCIS, with the exception of non-melanoma skin cancer (basal cell carcinoma and squamous cell carcinoma)
* Blood transfusions within the past 3 months
* Born biologically male

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Screening and Recall population. Women in the Screening Cohort would be consented just prior to a screening imaging session (within 3 months). Recruitment may also occur after a normal screening imaging session (within 3 months). Women in the Recall population include women called back for follow-up after abnormal imaging or clinical exam. Women at elevated risk of breast cancer development are included.
  The primary target population for recruitment is women at elevated risk (C or D breast density, family history, and/or genetic elevated risk) called back (recalled) for follow-up imaging or biopsy after an abnormal image with the following distribution: 60% White (non-hispanic), 14% Black, 18% Hispanic, 6% Asian and 2% other.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-10-27 (Estimated); Primary Completion 2027-06-14 (Estimated); Study Completion 2027-06-14 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 3 years
  Sensitivity (Se) if the test = TP/TP+FN), ratio of true positives to true positives and false negatives
Specificity | 3 years
  Specificity (Sp) of the test = TN/ (TN+FP), ratio of true negatives to the true negatives and false positives

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Vincere Cancer Center, Phoenix, Arizona
  - Weill Cornell Medicine of Cornell University, New York, New York
- Alberta Cancer Research Biobank, Calgary, Alberta, Canada
- Manchester University NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
This is not an interventional study.